CLINICAL TRIAL: NCT06471231
Title: Renal Outcomes in the Early Use of Vasopressin in the Treatment of Septic Shock
Acronym: EVSS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23171 - EVSS
Record Dates: First submitted 2024-05-14; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-05

CONDITIONS: Septic Shock; Renal Function Replacement
Keywords: vasopressin; norepinephrine; renal function replacement; Septic Shock
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus

STUDY DESIGN:
Intervention Model Description: Patients will be divided and randomized in a 1:1 ratio through a computer-generated scheme, when the dose of norepinephrine administered is ≥ 0.25 mcg/kg/min, into the following groups:
  * Group A: when the norepinephrine dosage is equal to or greater than 0.25 mcg/kg/min in the absence of adequate MAP (Mean arterial pressure >65 mmhg), vasopressin infusion will be associated with the standard dosage of 0.3UI/min.
  * Group B (control): the infusion of vasopressin at a dosage of 0.3 IU/min will be associated if norepinephrine exceeds the dosage of 0.5 mcg/kg/min in the absence of adequate MAP.
Who Masked: Investigator
Masking Description: An expert nephrology consultant has been included among the investigators to assess the need for CRRT according to KDIGO criteria, and he will be blinded to the subject allocation. In addition, the physicians who will perform ultrasound evaluation will be blinded to the subject allocation, in order to reduce the potential bias of overestimating the efficacy of the study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A: when the norepinephrine dosage is equal to or greater than 0.25 mcg/kg/min in the absence of adequate MAP (Mean arterial pressure >65 mmhg), vasopressin infusion will be associated with the standard dosage of 0.3UI/min.
  Interventions: Drug: vasopressin infusion when the norepinephrine dosage is equal to or greater than 0.25 mcg/kg/min
- Group B (Active Comparator): Group B (control): the infusion of vasopressin at a dosage of 0.3 IU/min will be associated if norepinephrine exceeds the dosage of 0.5 mcg/kg/min in the absence of adequate MAP.
  Interventions: Drug: vasopressin infusion when the norepinephrine dosage is equal to or greater than 0.5 mcg/kg/min

INTERVENTIONS:
Drug: vasopressin infusion when the norepinephrine dosage is equal to or greater than 0.25 mcg/kg/min — when the norepinephrine dosage is equal to or greater than 0.25 mcg/kg/min in the absence of adequate MAP (Mean arterial pressure >65 mmhg), vasopressin infusion will be associated with the standard dosage of 0.3UI/min.
  Arms: Group A
Drug: vasopressin infusion when the norepinephrine dosage is equal to or greater than 0.5 mcg/kg/min — the infusion of vasopressin at a dosage of 0.3 IU/min will be associated if norepinephrine exceeds the dosage of 0.5 mcg/kg/min in the absence of adequate MAP
  Arms: Group B

SUMMARY:
The aim of the present study is to verify whether the earlier association of vasopressin and norepinephrine, in patients in septic shock, determines variations in terms of use of renal function replacement techniques in the first 7 days of hospitalization in Intensive Care, compared to patients in whom vasopressin is added only when norepinephrine reaches a higher dose.

DETAILED DESCRIPTION:
The aim of the present study is to verify whether the earlier association of vasopressin and norepinephrine, in patients in septic shock, determines variations in terms of use of renal function replacement techniques in the first 7 days of hospitalization in Intensive Care, compared to patients in whom vasopressin is added only when norepinephrine reaches a higher dose. The study is aimed at patients admitted to the ICU with a diagnosis of septic shock on admission or in the first 24 hours of admission.

Patients will be divided and randomized in a 1:1 ratio through a computer-generated scheme, when the dose of norepinephrine administered is ≥ 0.25 mcg/kg/min, into the following groups:

* Group A: when the norepinephrine dosage is equal to or greater than 0.25 mcg/kg/min in the absence of adequate MAP (Mean arterial pressure >65 mmhg), vasopressin infusion will be associated with the standard dosage of 0.3UI/min.
* Group B (control): the infusion of vasopressin at a dosage of 0.3 IU/min will be associated if norepinephrine exceeds the dosage of 0.5 mcg/kg/min in the absence of adequate MAP.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from septic shock hospitalized in an intensive setting
* patients over 18 years and under 80 years of age
* patients within 24 hours of clinical diagnosis, and requiring, in this time window, a norepinephrine dosage equal to or greater than 0.25 mcg/kg/min according to the patient's ideal weight (IBW)
* patients capable of expressing informed consent to treatment.

Exclusion Criteria:

* patients in the absence of consent to participate in the study and to the processing of personal and particular data;
* patients under 18 years of age or over 80 years of age;
* patients who died within the first 24 hours of admission to the ICU;
* patients requiring a norepinephrine dosage lower than 0.25 mcg/kg/min in the first 24 hours of hospitalization in the ICU;
* patients with recent acute coronary syndrome (within the previous 7 days);
* patients with allergy/intolerance to the drugs used in the study or to any component of the study drug including excipients;
* pregnant patients;
* breastfeeding individuals;
* patients who need to start renal replacement treatment within 24 hours of admission to the ICU for dialysis emergencies that cannot be deferred;
* patients with a history of end-stage renal failure or already undergoing dialysis treatment (CKD stages 4 and 5, with glomerular filtration < 30 ml/min);
* single kidney patients;
* patients with bilateral renal hypoplasia;
* patients undergoing kidney transplant;
* patients undergoing haemoperfusion with an adsorbent cartridge for bacterial endotoxin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
30% or more reduction in terms of the use of renal function replacement | 7 days
  The primary objective of the study is to verify whether the earlier association of vasopressin and norepinephrine determines a 30% or more reduction in terms of the use of renal function replacement techniques in the first 7 days of hospitalization in the Intensive Care Unit (ICU), compared to patients in whom the vasopressin is added only when norepinephrine reaches a higher dosage.

SECONDARY OUTCOMES:
early association of vasopressin improves renal function | 7 days
  To assess the protective effect of early vasopressin association, the Kidigo score will be calculated for every subject at enrollment time, and daily, for 7 days. The maximum value and the greatest increase will be evaluated and compared between study and control group
rly addition of vasopressin modifies renal perfusion | 7 days
  verify whether the early addition of vasopressin modifies renal perfusion assessed ultrasoundally according to the CEUS method;
addition of vasopressin modifies the fluid balance of patients | 48 and 72 hours
  To assess the impact of early vasopressin association on the total amount of fluids administrated in the resuscitative phase of septic shock treatment, the fluid balance at 48 hours and 72 hours since ICU admission will be calculated for every subject, and compared between study and control group.
early combined treatment with vasopressin reduces the duration of the need for CRRT | 7 days
  verify whether early combined treatment with vasopressin reduces the duration of the need for CRRT (Continuous Renal Replacement Therapy) in patients who require such support during hospitalization in the ICU
early association of vasopressin reduces the onset of supraventricular arrhythmias | 7 days
  verify whether the early association of vasopressin reduces the onset of supraventricular arrhythmias (atrial fibrillation, atrial flutter, paroxysmal supraventricular tachycardia) during treatment with vasopressor drugs
intestinal and/or digital and/or limb ischemia; | 7 days since enrollment
  The incidence of intestinal and/or digital and/or limb ischemia during the study period (7 days since enrollment) will be evaluated and compared between study and control group.
Length of stay in ICU | 28 and 90 days
  Length of stay in ICU (days) will be compared between study and control group
Mortality | 28 and 90 days
  Mortality at 28 and 90 days will be evaluated for every subject and between study and control group

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Unità Sanitaria Locale, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided